CLINICAL TRIAL: NCT05147298
Title: Multilevel Physical Activity Intervention for Low Income Public Housing Residents
Brief Title: Community Walks: Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: H-42219; 1R01MD015165-01A1 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Physical Inactivity
Keywords: Public housing developments (PHDs); Environmental level interventions; Individual level interventions; eHealth phone program; Healthy living advocates
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Environmental group intervention (E only) (Experimental): Changing the environment surrounding the PHDs making it more amenable to walking and advocating for changes to the built environment
  Interventions: Other: Environment program
- Individual-level eHealth phone program intervention (I only) (Experimental): An automated telephone-based physical activity program.
  Interventions: Other: eHealth phone program
- Combined group (E and I interventions) (Experimental): Changing the environment surrounding the PHDs making it more amenable to walking and advocating for changes to the built environment and an automated telephone-based physical activity program.
  Interventions: Other: eHealth phone program; Other: Environment program
- Control group (no interventions) (No Intervention): No interventions for residents to increase activity levels.

INTERVENTIONS:
Other: eHealth phone program — The automated eHealth phone program uses text to speech technology to deliver educational content to increase awareness, confidence, and motivation for physical activity.
  Arms: Combined group (E and I interventions); Individual-level eHealth phone program intervention (I only)
Other: Environment program — The environment surrounding the PHDs will be changed to make it more amenable to walking by creating walking trails and walking maps and using Healthy Living Advocates (HLA)-led walking groups within the community. Also advocating for changes to the built environment.
  Arms: Combined group (E and I interventions); Environmental group intervention (E only)

SUMMARY:
This research study will investigate the independent effects of an environmental intervention (E only), an individual-level eHealth phone program intervention (I only), or both (E+I) on changes in moderate intensity physical activity. A cluster randomized design will be implemented whereby all residents of one of 12 of Boston's public housing developments (PHDs) will be randomized to one of the four study groups (E only, I only, E+I, or control). The activities with this multilevel design include:

* Screening/enrollment/baseline assessment activities
* Environmental components to promote moderate intensity walking and other physical activity at the PHDs
* Changing the environment surrounding the development making it more amenable to walking through the creation of walking trails and walking maps; and advocating for changes to the built environment
* Healthy Living Advocates (HLA)-led walking groups within the community
* Individual level components to increase motivation and self-efficacy for physical activity
* eHealth program, an automated telephone-based physical activity program
* 12-month and 24-month follow up assessment activities

The investigators hypothesize that the participants living in the PHDs in any of the three intervention groups (E only, I only, and E+I combined) will increase minutes of moderate intensity physical activity more than participants in control group developments at 24-month follow up. It is further expected that delivery of an intervention package targeting environmental and social cues to become active, combined with an individual level intervention, will improve overall physical activity levels to recommended guidelines at the development level. The findings will inform future health promotion efforts among residents in public housing developments.

ELIGIBILITY:
Inclusion Criteria:

* Willing to wear device to track physical activity during assessment periods
* Able to speak English or Spanish
* Current resident of Boston Public Housing Development or housing property on Boston Housing Authority owned land
* No plans to move within the next 2 years
* Has access to a phone (of any kind)

Exclusion Criteria:

* Currently enrolled in a research study about physical activity that is incompatible with study participation
* Unable to provide informed consent in judgement of research assistant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in minutes of light, moderate, and vigorous intensity physical activity per day at 12 months | baseline, 12 months
  Assessed by (1) evaluating the proportion of accelerometers distributed and returned, (2) downloading the data from the devices, (3) processing the data (e.g., removing outliers), and (4) examining the proportion that have valid data (i.e., minimum 3 days of wear).
Change in minutes of light, moderate, and vigorous intensity physical activity per day at 24 months | baseline, 24 months
  Assessed by (1) evaluating the proportion of accelerometers distributed and returned, (2) downloading the data from the devices, (3) processing the data (e.g., removing outliers), and (4) examining the proportion that have valid data (i.e., minimum 3 days of wear).

SECONDARY OUTCOMES:
Evaluate the mediator effects of motivation | baseline, 12 months, 24 months
  This outcome will be assessed by analyzing participants' responses to relevant questions in an Investigator developed questionnaire.
Evaluate the mediator effects of self-efficacy | baseline, 12 months, 24 months
  This outcome will be assessed by analyzing participants' responses to relevant questions in an Investigator developed questionnaire.
Evaluate the mediator effects of neighborhood walkability | baseline, 12 months, 24 months
  This outcome will be assessed by analyzing participants' responses to relevant questions in an Investigator developed questionnaire.
Evaluate the mediator effects of support from HLAs | baseline, 12 months, 24 months
  This outcome will be assessed by analyzing participants' responses to relevant questions in an Investigator developed questionnaire.
Evaluate the mediator effects fidelity to the interventions | baseline, 12 months, 24 months
  This outcome will be assessed by analyzing participants' responses to relevant questions in an Investigator developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Quintiliani, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quintiliani LM, Dedier J, Amezquita M, Sierra-Ruiz M, Romero D, Murillo J, Mahar S, Goodman M, Kane JB, Cummings D, Woolley TG, Spinola I, Crouter SE. Community Walks: a cluster randomized controlled trial of a multilevel physical activity intervention for low income public housing residents. BMC Public Health. 2023 Aug 31;23(1):1676. doi: 10.1186/s12889-023-16574-y. PMID 37653386